CLINICAL TRIAL: NCT01223118
Title: Evaluation of the Impact of Vitrification on the Reproductive Performance and Potential of Human Oocytes
Brief Title: Evaluation of the Impact of Vitrification on Oocytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RMA-2010-02
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Fertilization
Keywords: Oocyte; vitrification; IVF; PGD; embryo biopsy
MeSH Terms: interventions — Vitrification; Prostaglandins D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oocyte Vitrification (Experimental): Each patient will have oocytes randomized into two groups immediately after retrieval. Half of oocytes will be vitrified, thawed and inseminated. The other half will be inseminated only. All embryos will be biopsied for PGD prior to transfer and one embryo from each group will be transferred (vitrification and control groups). Following delivery, buccal swabs will be collected on all infants.
  Interventions: Procedure: Vitrification and PGD

INTERVENTIONS:
Procedure: Vitrification and PGD — Half of the oocytes retrieved from each patient will undergo vitrification, immediate thaw and insemination. All embryos will undergo biopsy for PGD prior to transfer.
  Other Names: Vitrification; PGD

SUMMARY:
The purpose of this study is to determine the rate of cryosurvival of mature oocytes following vitrification, and to then compare the reproductive potential of vitrified oocytes relative to those which have not been cryopreserved.

DETAILED DESCRIPTION:
This study will recruit patients from the NY/NJ/CT/eastern PA area only.

Cryopreservation of human oocytes has a great potential to preserve or extend fertility in the face of disease whose treatment would result in a loss of ovarian function. (malignancy, severe autoimmune disease, etc.). It would also provide a means of quarantining oocytes to be used in oocyte donation to provide the lowest possible risk of infection.

There are two methods for storage of oocytes: slow freezing or vitrification. Slow freezing is the conventional method and has been successfully used for embryos since 1983 and more recently for oocytes. Recent reports indicate that vitrification may be more successful than slow freezing. However, the technique has not been rigorously validated to date. The aim of this study is to determine the rate of cryosurvival of mature oocytes following vitrification, and to then compare the reproductive potential of vitrified oocytes relative to those which have not been cryopreserved.

Patients will undergo ovarian stimulation for in vitro fertilization (IVF) according to the protocol recommended by their primary doctor. After retrieval, mature oocytes will be divided in half. One half will undergo vitrification, immediate thaw and intracytoplasmic sperm injection (ICSI). The other half will undergo just ICSI. All embryos will then develop on identical culture until day 3 or day 5. Prior to transfer, the best embryo from each group will undergo biopsy for genetic fingerprinting. The patient will have a 2 embryo transfer (one from each group). All extra embryos will be biopsied for pre-implantation genetic diagnosis (PGD) prior to being cryopreserved. If the patient becomes pregnant, we will follow up with an additional blood draw at approximately 9 weeks gestation and buccal swabs after the delivery of the infant(s).

ELIGIBILITY:
This study will recruit patients from the NY/NJ/CT/eastern PA area only.

Inclusion Criteria:

1. No prior failed IVF treatment cycle
2. Female partner less than 35 years of age at time of onset of the IVF cycle
3. Normal maximum prior day 3 follicle stimulating hormone (FSH) level (< or = 10 IU/L)
4. Total basal antral follicle count greater than or equal to 12
5. Male partner with greater than 100,000 total motile spermatozoa Donor sperm is acceptable but the couples will be required to provide one additional vial for DNA analysis
6. Body Mass Index (BMI) ≤ 32 kg/m2

Exclusion Criteria:

1. Diagnosis of chronic oligoovulation or anovulation (cycle typically occurring less often than every 38 days)
2. Diagnosis of endometrial insufficiency
3. Clinical indication for PGD (undergoing IVF with PGD to rule out a known genetic defect)
4. Use of testicular aspiration or biopsy procedures to obtain sperm
5. Unevaluated ovarian mass
6. Presence of hydrosalpinges which communicate with the endometrial cavity
7. Any contraindication to undergoing in vitro fertilization or gonadotropin stimulation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Aneuploidy Rate (evaluation of whether embryo is chromosomally normal) | 1 year
  Compare the rate of chromosomally-abnormal embryos among embryos originating from vitrified oocytes versus embryos originating from fresh/control oocytes.

SECONDARY OUTCOMES:
Delivery rates | 1 year
  All embryos will be biopsied prior to transfer and DNA samples will be collected from all infants. Compare embryonic and infant DNA to evaluate whether the live birth resulted from a vitrified or a fresh/control oocyte.
Paired Sustained Implantation Rate (number of viable fetuses beyond the first trimester per embryo transferred) | 1 year
  Among patients with a paired two blastocyst transfer, compare the implantation rate of embryos originating from vitrified oocytes versus embryos originating from fresh/control oocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- United States (2):
  - Reproductive Medicine Associates of New Jersey, Morristown, New Jersey
  - Reproductive Medicine Assoicates of PA at Lehigh Valley, Allentown, Pennsylvania